CLINICAL TRIAL: NCT00246753
Title: A Phase II Study of Oral Once Daily GW572016 (Lapatinib) In Patients With Hormone Refractory Prostate Cancer
Brief Title: Lapatinib in Treating Patients With Prostate Cancer That Did Not Respond to Hormone Therapy
Acronym: NRR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0505; CDR0000550151 (Other: PDQ number)
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Trial (Other): Single Arm Trial where each patient receives GW572016 (lapatinib ditosylate) at a dose of 1500mg daily initially until disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate

INTERVENTIONS:
Drug: lapatinib ditosylate — 1500 mg, daily until disease progression
  Other Names: GW572016

SUMMARY:
RATIONALE: Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well lapatinib works in treating patients with prostate cancer that did not respond to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the proportion of patients with hormone-refractory prostate cancer who experience > 50% decline in prostate-specific antigen (PSA) after treatment with lapatinib ditosylate.

Secondary

* Determine the safety of this drug in these patients.
* Determine the time to PSA progression in patients treated with this drug.
* Determine the molecular correlates and predictive biomarkers of response in patients treated with this drug.

OUTLINE: This is a multicenter, open-label study.

Patients receive oral lapatinib ditosylate once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Serum samples are collected for biomarker analysis at baseline and every 4 weeks.

After completion of study treatment, patients are followed at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of adenocarcinoma of the prostate.
* On androgen deprivation therapy for prostate cancer (either bilateral orchiectomy or medical castration with the testosterone level of <50 ng/dl)
* Biochemical progression on androgen deprivation therapy with minimum PSA of 5 ng/ml. Progression is defined as two successive rises in PSA, measured at least one week apart. See section 4.1 for additional criteria.
* Minimum of 4-6 weeks off anti-androgen therapy (4 weeks for flutamide, 6 weeks for bicalutamide and nilutamide).
* Minimum of 4 weeks off other hormonal therapy (i.e. ketoconazole, megestrol acetate, aminoglutethimide)
* Minimum of 4 weeks from any prior radiation therapy, surgery, chemotherapy or other investigational agent.
* Patients must discontinue use of any herbal supplements prior to study initiation.
* No prior or concurrent exposure to cytotoxic chemotherapy.
* Age > 18 years.
* Life expectancy greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram or multigated acquisition scan (MUGA) scan.
* Men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation since the effects of GW572016 on the developing human fetus at the recommended therapeutic dose are unknown.
* Ability to swallow and retain oral medication.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had prior treatment with ErbB family targeting therapies.
* Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Prior chemotherapy for prostate cancer
* Patients with known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GW572016.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* A history of a positive HIV test in the past.
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
* Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors (please refer to section 3.2.2 for a list of medications).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-10; Primary Completion 2012-07 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young Whang, MD, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00246753?term=LCCC0505&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men with castration-resistant prostate cancer were recruited from 3 local institutions from 11/11/2005 to 8/29/2007.
Pre-assignment Details: Of the 35 patients initially recruited, 4 were not eligible. One patient was removed in order to receive more aggressive treatment and another patient was removed due to disease progression or death prior to protocol therapy. 29 patients were enrolled.
Groups:
- Single Arm Trial: Single Arm Trial
  lapatinib ditosylate: 1500 mg, daily until disease progression
Period: Overall Study
Arm/Group | Single Arm Trial
Started | 29
Completed | 21
Not Completed | 8
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2
Not completed — Adverse Event | 2
Not completed — Unacceptable toxicity | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 72.5 [58 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29
PSA [Median (Full Range); unit: ng/mL] — Prostate-specific antigen, or PSA, is a protein produced by cells of the prostate gland. The PSA test measures the level of PSA in an individual's blood.The results are usually reported as nanograms of PSA per (ng/mL) of blood. In this study PSA response is defined as >50% decrease in PSA from baseline for 2 successive measurements at lease 4 weeks apart.
  ng/mL | 21.6 [4.5 to 196.5]
Alkaline phosphatase [Median (Full Range); unit: U/L] — Alkaline phosphatase (ALP) is an enzyme found in your bloodstream. ALP helps break down proteins in the body and exists in different forms, depending on where it originates. Normal range is 44 to 147 U/L ( units per liter)
  U/L | 85 [55 to 110]
Hemoglobin [Median (Full Range); unit: grams per deciliter] — Hemoglobin is a component of red blood cells. The normal level is around 15 grams per deciliter (g/dl) and lower levels in men with prostate cancer indicate a worse prognosis.
  grams per deciliter | 13 [11 to 14.7]
Disease Status [Count of Participants; unit: Participants] — Metastasis is the development of secondary malignant growths at a distance from a primary site of cancer. Measurable disease is the presence of at least one measurable lesion. This is based on RECIST criteria. Response Evaluation Criteria In Solid Tumors (RECIST) is a set of published rules that defines the status of cancer in a patient. Looking at when tumors improve, stay the same, or worsen.
  Participants
    Bone metastases only | 8
    Measurable disease only | 7
    Both bone and measureable disease | 7
    No metastasis | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Decline in Prostate-specific Antigen
Description: Determine the number of patients with hormone-refractory prostate cancer who experience > 50% decline in PSA from baseline for 2 successive measurements at least 4 weeks apart after treatment with lapatinib ditosylate.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 21
Participants | 2

2. Secondary Outcome: Time to Prostate-Specific Antigen (PSA) Progression
Description: Measured from start date of treatment to date of PSA progression, defined as a 25% increase above the pretreatment value or the nadir PSA (whichever is lower) and a minimum increase of 5 ng/ml, confirmed 2 or more weeks later.
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 21
days | 29 [29 to 56]

3. Secondary Outcome: Predictive Molecular Markers of Response to Treatment With Lapatinib (GW572016)
Description: To assess the correlation between expression of molecular markers and patient response to treatment with GW572016
Time Frame: 4 years
Population: Data were not collected.
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Single Arm Trial
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 4/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Trial (N=29)
Epigastric pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Trial (N=29)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2
Alkaline phosphatase (Metabolism and nutrition disorders) | 1
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 3
Anorexia (Gastrointestinal disorders) | 9
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1
Hearing loss (Ear and labyrinth disorders) | 1
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1
Bladder spasms (Renal and urinary disorders) | 2
Elevated Phosphorus (Blood and lymphatic system disorders) | 1
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Creatinine (Investigations) | 3
Dehydration (Gastrointestinal disorders) | 1
Skin lesions (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 22
Distension/bloating, abdominal (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 2
Dry eye syndrome (Eye disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Edema: limb (General disorders) | 5
Fatigue (asthenia, lethargy, malaise) (General disorders) | 21
Flatulence (Gastrointestinal disorders) | 4
Flu-like syndrome (General disorders) | 4
Epigastric pain (Gastrointestinal disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 8
Hemoglobin (Blood and lymphatic system disorders) | 12
Hemorrhage, GU - Bladder (Renal and urinary disorders) | 1
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1
Gross hematuria (Vascular disorders) | 1 — 1 x daily
Hot flashes/flushes (Vascular disorders) | 1
Hypertension (Cardiac disorders) | 2
Incontinence, urinary (Renal and urinary disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Appendix (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 3
Insomnia (Psychiatric disorders) | 3
Joint-function (Musculoskeletal and connective tissue disorders) | 1
Leak (including anastomotic), GU - Bladder (Renal and urinary disorders) | 1
Leukocytes (total WBC) (Investigations) | 1
Lymphopenia (Investigations) | 6
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 5
Memory impairment (Nervous system disorders) | 2
Mucositis/stomatitis (clinical exam) - Anus (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 2
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Right-sided (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 3
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Neuropathy: sensory (Nervous system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Obstruction, GU - Bladder (Renal and urinary disorders) | 1
Conjunctivitis (Eye disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 3
Pain - Cardiac/heart (Cardiac disorders) | 1
Pain - Chest wall (General disorders) | 2
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 3
Pain - Head/headache (Nervous system disorders) | 5
Pain - Joint (Musculoskeletal and connective tissue disorders) | 5
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1
Shoulder Pain (General disorders) | 3
Pain - Pain NOS (General disorders) | 1
Pain-Stomach (Gastrointestinal disorders) | 1
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 7
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3
Lower urinary tract symptoms (Renal and urinary disorders) | 1
Rigors/chills (General disorders) | 2
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1
Taste alteration (dysgeusia) (Nervous system disorders) | 2
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1
Tremor (Nervous system disorders) | 2
Urinary frequency/urgency (Renal and urinary disorders) | 5
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Weight loss (Investigations) | 3
Oily skin (Skin and subcutaneous tissue disorders) | 1
Bleeding mole (Skin and subcutaneous tissue disorders) | 1
Heel pain (General disorders) | 3
Dysuria (Renal and urinary disorders) | 1
Large stools (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days